CLINICAL TRIAL: NCT01516918
Title: A Multicenter, Open-Label Phase 2b Pilot Study to Evaluate the Efficacy and Safety of Quadruple Therapy (VX-222, Telaprevir, Peginterferon-Alfa-2, and Ribavirin) in Subjects With Genotype 1 Chronic Hepatitis C With Compensated Cirrhosis
Brief Title: A Study to Evaluate the Efficacy and Safety of Quadruple Therapy (VX-222, Telaprevir,Peginterferon-Alfa-2a, Ribavirin) in Subjects With Chronic Hepatitis C With Compensated Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX11-222-106
Record Dates: First submitted 2012-01-13; First posted 2012-01-25 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — lomibuvir; telaprevir; Ribavirin; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Quadruple Regimen (Experimental): All subjects will receive active study drugs (quadruple regimen: VX-222, telaprevir,Peg-IFN, and RBV) for a fixed treatment duration of 24 weeks.
  Interventions: Drug: VX-222; Drug: telaprevir; Drug: ribavirin; Biological: peginterferon-alfa-2a

INTERVENTIONS:
Drug: VX-222 — tablet, 400-mg twice daily
Drug: telaprevir — tablet, 1125-mg twice daily
  Other Names: Incivek, VX-950, Incivo
Drug: ribavirin — tablet, 1000-mg per day for subjects weighing <75 kg and 1200 mg per day for subjects weighing ≥75 kg, twice daily
  Other Names: Copegus
Biological: peginterferon-alfa-2a — subcutaneous injection, 180-mcg, once weekly
  Other Names: Pegasys

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of a quadruple regimen (VX-222, telaprevir, pegylated interferon, and ribavirin)in subjects with hepatitis C with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have genotype 1 Chronic Hepatitis C
* Subjects must have compensated cirrhosis
* Subjects may either be treatment naïve, or may have received a course of Peg IFN/RBV without evidence of response. Subjects who are considered to be relapsers to Peg IFN/RBV, or who are partial or null responders will be considered
* Subjects with hemophilia may be permitted to enroll with permission of the medical monitor

Exclusion Criteria:

* Any previous treatment with an investigational drug or drug regimen for the treatment of hepatitis C, or previous treatment with an approved protease inhibitor
* Any contraindication to Peg-IFN or RBV therapy
* Evidence of hepatic decompensation: history of ascites, hepatic encephalopathy, or bleeding esophageal varices
* A history of acquired immunodeficiency infection, organ transplantation or have an ongoing requirement for immunosuppressive medicines

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2012-02; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who have a sustained virologic response at 12 weeks after the last planned dose of treatment (SVR12) | 12 weeks

SECONDARY OUTCOMES:
The safety and tolerability as assessed by adverse events, vital signs, 12-lead electrocardiograms and laboratory assessments. | up to 48 weeks
The proportion of subjects who have an SVR 24 weeks after the last planned dose of the study drug (SVR24) | 24 weeks
The proportion of subjects who achieve undetectable HCV RNA at Weeks 2, 4, 8, and 12 after the first dose of study drug, and at the end of planned study drug treatment | up to week 12
The proportion of subjects who have on-treatment virologic failure defined as subjects who either meet a futility rule or who complete the assigned treatment duration and have HCV RNA at the end of study drug treatment | up to 48 weeks
The association of the IL-28B genotype with SVR12 | 12 weeks
  Proportion of subjects who have SVR12 by IL-28B genotype
The amino acid sequence of the nonstructural (NS)3 and NS5B proteins in subjects who have treatment failure | After the last planned dose of study drug or after time of failure
  The identity and observed frequency of viral variants as compared to wild-type virus will be measured.
VX-222, telaprevir, and RBV plasma concentrations and Peg-IFN serum concentrations | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (43):
- United States (28):
  - Birmingham, Alabama
  - San Diego, California
  - Englewood, Colorado
  - Bradenton, Florida
  - Jacksonville, Florida
  - Tampa, Florida
  - Marietta, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Boston, Massachusetts
  - Detroit, Michigan
  - Lebanon, New Hampshire
  - Egg Harbor, New Jersey
  - Manhasset, New York
  - New York, New York
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Providence, Rhode Island
  - Germantown, Tennessee
  - Arlington, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (3):
  - Vancouver, British Columbia
  - London, Ontario
  - Montreal, Quebec
- Germany (6):
  - Cologne
  - Hamburg
  - Heidelberg
  - Hessen
  - Saschen
  - Stuttgart
- Poland (3):
  - Bialystok
  - Mysłowice
  - Wroclaw
- United Kingdom (3):
  - London
  - Plymouth
  - Scotland